CLINICAL TRIAL: NCT03239288
Title: A Randomized, Controlled, Crossover Study to Assess the Glucose and Insulin Excursions of a Test Fiber
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cargill (Industry)
Collaborators: Biofortis Clinical Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: BIO-1706
Record Dates: First submitted 2017-08-01; First posted 2017-08-04 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Healthy
Keywords: Fiber; Postprandial glucose; Insulin; Resistant Starch Type 4
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, double-blind, crossover trial that includes one screening visit and two test visits separated by a washout period of 4-7 days. At Visit 1 (day -7), subjects will provide informed consent and undergo screening assessments. Test day instructions will also be provided.
  At Visit 2 (day 0), subjects will arrive at the clinic fasted (10-14 h, water only, anchored to the t = -15 min blood draw), to undergo clinic visit procedures. Eligible subjects will be randomly assigned to a randomization sequence and will undergo the glycemic and insulinemic response test with blood glucose concentrations assessed via capillary measurement and insulin concentrations assessed via venous measurement.
  At Visit 3 (day 7), subjects will return to the clinic for clinic visit procedures. Subjects will then crossover to the next study product in their test sequence and repeat the glycemic/insulinemic response test described above for Visit 2.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control digestible carbohydrate (Placebo Comparator): Control baked breakfast bar
  Interventions: Other: Control digestible carbohydrate
- Test resistant starch type 4 (Experimental): Test baked breakfast bar
  Interventions: Other: Test resistant starch type 4

INTERVENTIONS:
Other: Control digestible carbohydrate — Single serving of control product
  Arms: Control digestible carbohydrate
Other: Test resistant starch type 4 — Single serving of test product
  Arms: Test resistant starch type 4

SUMMARY:
The objective of this trial is to evaluate the postprandial glucose and insulin responses to replacing digestible carbohydrates with resistant starch type 4 (RS4) in a baked product in healthy men and women. A randomized, double-blinded cross-over study will be conducted comparing two foods (a reference food and a test food). The primary outcome variable will be the incremental area under the curve (iAUC) for capillary glucose from pre-product consumption (average of t = -15 and -5 min) to 120 min (iAUC0-120 min). This study will provide substantiation for a beneficial reduction in glycemic response followed by the consumption of the active product containing an efficacious dose of resistant starch type 4 (RS4).

DETAILED DESCRIPTION:
The study is a randomized, controlled, double-blind, crossover trial that includes one screening visit (Visit 1; day -7) and two test visits (Visits 2 and 3; days 0 and 7) which are separated by a washout period of 4-7 days. At Visit 1 (day -7), subjects will provide informed consent and undergo screening assessments including evaluations of medical history, prior/current medication/supplement use, inclusion and exclusion criteria, height, body weight, BMI, vital signs, and Vein Access Scale. A fasting capillary blood glucose will be assessed for eligibility purposes and an in-clinic urine pregnancy test (all women) will also be obtained. Subjects will then be dispensed a 24-h Diet Record with instructions to record intake the day prior to Visit 2 (day 0). At Visit 2 (day 0), subjects will arrive at the clinic fasted (10-14 h, water only, anchored to the t = -15 min blood draw), to undergo clinic visit procedures. Adverse events (AE) will be assessed and subjects will be queried about test day instructions compliance. Additionally, the 24-h Diet Record will be collected and reviewed. Eligible subjects will be randomly assigned to a randomization sequence and will undergo the glycemic and insulinemic response test with blood glucose concentrations assessed via capillary measurement and insulin concentrations assessed via venous measurement. Blood samples (capillary and venous) will be obtained at t = -15 and -5 ± 5 min. Subjects will consume the study product in its entirety within 10 min at t = 0 min with 8 oz of water. Capillary and venous blood samples will be obtained at t = 15, 30, 45, 60, 90, and 120 ± 5 min, where t = 0 min is the start of study product consumption, to assess glucose and insulin concentrations. Subjects will be provided one-8 oz bottle of water to consume at t = 0 to 60 min and one-8 oz bottle of water to consume at t = 61 to 120 min. Water consumption will be recorded and replicated at the subsequent test visits. AEs will be assessed and subjects will be dispensed a blank/new 24-h Diet Record to record all food and beverage consumed the day prior to Visit 3, day 7; as well as a copy of the completed 24-h Diet Record (from day -1) with instructions to replicate the same food and beverage intake as closely as possible the day prior to the next test visit (Visit 3, day 7). Test day instructions will also be provided. At Visit 3 (day 7), subjects will return to the clinic for clinic visit procedures. AEs will be assessed and subjects will be queried about test day instructions compliance. The 24-h Diet Record will be collected and study staff will review the 24-h Diet Record to compare food and beverage consumption to the day -1 Diet Record for consistency. Subjects will then crossover to the next study product in their test sequence and repeat the glycemic/insulinemic response test described above for Visit 2. At the conclusion of the glycemic/insulinemic response test, AEs will be assessed.

An evaluable sample size of 19 is required to observe a statistically significant difference between active and control products (α = 0.05 (2- tailed); power = 80%) assuming that the glucose response of the Cargill active product is 61% of that of the control product and standard deviation is 65% of the mean value (standard deviation estimation is based on a recently completed proprietary study conducted by Biofortis on baked products containing different amounts of fiber). To account for possible attrition, a total of 22 subjects will be enrolled. Each subject will consume a single serving of the control or active product. These consumption events will be separated by at least 4 days.

All statistical analyses will be conducted using Statistical Analysis Systems (SAS) for Windows (version 9.4, Cary, NC) and/or R 3.3.1 (R Core Team 2016). The data will be analyzed for the modified intent-to-treat population, which will include all subjects who complete the test condition and the reference product. Assessment for outliers, as per the International Organization for Standardization (ISO) standards, will also be conducted. All decisions regarding subject population and data inclusion will be documented prior to database lock. Descriptive statistics [number of subjects, mean, standard deviation, standard error of the mean (SEM), median, interquartile limits, minimum and maximum or frequency counts] will be presented for subject demographics and anthropometric measurements collected at screening/baseline. Incremental area under the curve (iAUC) 0-120 min will be calculated as outlined in ISO 26642:2010(E) for each subject. Descriptive statistics (i.e. number of subjects, minimum and maximum, median, inter-quartile limits, mean, SEM, and standard deviation) will be presented for all the continuous outcomes for each test group. All tests of significance, unless otherwise stated, will be performed at alpha=0.05, two sided. A repeated measures analysis of covariance (ANCOVA) will be used to assess differences between test groups for the primary and secondary outcome variables with the exception of the comparisons between groups for glucose and insulin concentrations at each time point. Initial repeated measures ANCOVA models will contain terms for test group, test sequence, and test period, with test group specified as a repeated effect and subject nested within sequence. Models will be reduced using a backward selection method until only significant terms or test group remains in the model. Appropriate least squares mean values and corresponding SEM will be derived from the final model for each test group. Assumption of normality of residuals will be investigated at the 5% level with the Shapiro-Wilk test (Shapiro 1965). If the normality assumption is not satisfied, then an analysis based on ranks will be performed. Average blood glucose response curve, as described in ISO 26642:2010(E), and time curve plots of the observed glucose and insulin concentration per time point per test product will be presented. Glucose concentrations will be provided in mg/dL and insulin concentrations will be provided at μIU/mL.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a generally healthy male or female, 20-45 years, inclusive.
* Body mass index (BMI) 18.5 to 27.0 kg/m2, inclusive, at Visit 1 (day -7).
* Subject has a rating of 7 to 10 on the Vein Access Scale at Visit 1 (day -7).
* If a smoker, subject has no plans to change smoking habits during the study period and is able to abstain from tobacco products at least 1 hour prior to and during each test visit.
* Normally active and judged by the Clinical Investigator/Medical Monitor to be in general good health on the basis of medical history.
* Willing to abstain from alcohol consumption and avoid vigorous physical activity for 24 hours prior to and during test visits.
* Subject is willing to maintain physical activity patterns, body weight, and habitual diet throughout the trial.
* Understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the Clinical Investigator/Medical Monitor.
* Subject has no health conditions that would prevent him/her from fulfilling the study requirements as judged by the Clinical Investigator/Medical Monitor on the basis of medical history and routine laboratory test results.
* Willing to maintain current use of vitamins, minerals, and other supplements throughout the trial. On test days, subject agrees not to take any vitamins, minerals, or other dietary supplements until dismissal from the clinic. Failure to comply will result in a rescheduled test visit.
* For females on oral contraceptives, the subject must be on a stable dose of oral contraceptives (defined as same dose for the past 90 d prior to Visit 1; day -7).

Exclusion Criteria:

* Fasting blood glucose ≥110 mg/dL at Visit 1 (day -7) or diagnosed diabetes mellitus. No retest will be allowed.
* History or presence of uncontrolled and/or clinically important pulmonary (including uncontrolled asthma), cardiac (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), hepatic, renal, gastrointestinal (including but not limited to inflammatory bowel diseases, such as Crohn's disease, ulcerative colitis, or other gastrointestinal conditions that may interfere with the absorption of the study product), endocrine, hematologic, immunologic, neurologic (such as Alzheimer's or Parkinson's disease), psychiatric (including depression and/or anxiety disorders) or biliary disorders.
* Subject has a history of bariatric surgery for weight reducing purposes.
* Subject has had a weight loss or gain >4.5 kg in the 3 months prior to Visit 1 (day -7).
* Subject has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg) at Visit 1 (day -7).
* History or presence of cancer in the prior two years, except for non-melanoma skin cancer.
* Subject has any signs or symptoms of an active infection of clinical relevance (e.g., urinary tract or respiratory) within 5 d prior to any test visit. If an infection occurs during the study period, test visits should be rescheduled until all signs and symptoms have resolved (at the discretion of the Clinical Investigator/Medical Monitor) and any intervention (e.g., antibiotic therapy) has been completed at least 5 d prior to testing.
* Has used medications known to influence carbohydrate metabolism, including, but not limited to, protease inhibitors, antipsychotics, adrenergic receptor blockers, diuretics, thiazolidinediones, metformin, and systemic corticosteroids, within 4 weeks of Visit 1 (stable doses of vitamin and mineral supplements are allowed).
* Subject has used weight-loss drugs (including over-the-counter medications and/or supplements) or programs within 4 weeks prior to Visit 1 (day -7).
* Subject has experienced any major trauma or surgical event within three months of Visit 1 (day -7).
* Recent (within 4 weeks of Visit 1) use of antibiotics.
* Recent history of (within 12 months of Visit 1) or strong potential for alcohol or substance abuse. Alcohol abuse define as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
* Subject has a known food allergy or intolerance, or sensitivity to any ingredients in the study products.
* Subject has extreme dietary habits (e.g., Atkins diet, very high protein, vegetarian), in the opinion of the Clinical Investigator/Medical Monitor.
* Subject is a female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the stable use of a medically approved form of contraception throughout the study period.
* Exposure to any non-registered drug product within 30 d prior to Visit 1 (day - 7).
* Individual has a condition the Clinical Investigator/Medical Monitor believes would interfere with his ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the subject at undue risk.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2017-07-28 (Actual); Study Completion 2017-07-28 (Actual)

PRIMARY OUTCOMES:
Incremental area under the curve (iAUC) for glucose | Capillary glucose test at t = -15 and -5 and at t = 15, 30, 45, 60, 90, and 120 min after product consumption
  Incremental area under the curve (iAUC) for capillary glucose across 2h

SECONDARY OUTCOMES:
Maximum concentration (Cmax) for glucose | 0-120 minutes
  Maximum concentration for capillary glucose within the tested time interval
Time to maximum concentration (tmax) for glucose | 0-120 minutes
  Time to maximum concentration for capillary glucose within the tested time interval
Incremental area under the curve (iAUC) for insulin | Venous insulin test at t = -15 and -5 and at t = 15, 30, 45, 60, 90, and 120 min after product consumption
  Incremental area under the curve (iAUC) for venous insulin across 2h
Maximum concentration (Cmax) for insulin | 0-120 minutes
  Maximum concentration for capillary venous insulin within the tested time interval
Time to maximum concentration (tmax) for insulin | 0-120 minutes
  Time to maximum concentration for venous insulin within the tested time

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Kelley, MD, Principal Investigator — Biofortis Clinical Research, Inc.
Locations (1):
- Biofortis Clinical Research, Addison, Illinois, United States

REFERENCES:
- [Derived] Mah E, Garcia-Campayo V, Liska D. Substitution of Corn Starch with Resistant Starch Type 4 in a Breakfast Bar Decreases Postprandial Glucose and Insulin Responses: A Randomized, Controlled, Crossover Study. Curr Dev Nutr. 2018 Aug 9;2(10):nzy066. doi: 10.1093/cdn/nzy066. eCollection 2018 Oct. PMID 30338311